CLINICAL TRIAL: NCT02145572
Title: Metabolomic Profiling in Adolescents With Obesity and Diabetes
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Dr Jane Kim, Associate Physician, Department of Pediatrics, University of California, San Diego
Other Study IDs: UCSD-IRB-140054
Record Dates: First submitted 2014-05-19; First posted 2014-05-23 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Metabolomics; Obesity; Diabetes; Diabetic Nephropathies
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obese adolescents with type 2 diabetes: No intervention
- Obese adolescents without diabetes: No intervention
- Healthy non-obese adolescents: No intervention

SUMMARY:
The purpose of this study is to identify unique metabolite signatures associated with the development of Type 2 diabetes and diabetic kidney disease in children.

We have a sub-study, with the purpose to validate the presence of a genetic marker (DENND1A) in the urine of adolescent females with polycystic ovarian syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Age of 13-19 years
* Gender: male and female
* Ethnic background: any
* Obesity will be defined as BMI >95th percentile for age/gender
* Diagnosis of diabetes will be defined by current American Diabetes Association criteria
* Diabetes duration < 2.5 years
* Absence of pancreatic autoimmunity (GAD65 and ICA512 and Insulin autoantibody)
* Adult caregiver willing to actively support study participation
* Signed parental informed consent form and adolescent assent form
* For PCOS substudy, the diagnosis of PCOS will be defined according to the 1990 US National Institute of Health (NIH) criteria (oligomenorrhea, clinical or biochemical signs of hyperandrogenism, and exclusion of other known disorders)

Exclusion Criteria:

* Creatinine clearance <60 mL/min (calculated from estimated GFR)
* Other significant organ system illness or condition (including psychiatric or developmental disorder) that, in the opinion of the investigator, would prevent participation.
* For PCOS substudy, use of medications that effect androgen levels in the blood (i.e. oral contraceptive pills, or metformin) for the last 3 months prior to enrollment

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be recruited from clinical practices affiliated with Rady Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-05; Primary Completion 2019-04 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Differences in metabolite concentrations measured by mass spectrometry, comparing blood and urine samples from obese adolescents with type 2 diabetes, obese adolescents without diabetes, and age-matched healthy non-obese controls. | 2 years

OTHER OUTCOMES:
Validation of presence of DENND1A isoform in the urine of adolescent females with polycystic ovarian syndrome | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jane J Kim, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Rady Children's Hospital, San Diego, California, United States